CLINICAL TRIAL: NCT01607593
Title: A Retrospective And Multicenter Survey To Investigate The Dosage, Efficacy And Safety Of Sertraline In Posttraumatic Stress Disorder Patients
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0501099
Record Dates: First submitted 2012-05-21; First posted 2012-05-30 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Retrospective; Sertraline; Posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sertraline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sertraline (Zoloft)
  Interventions: Drug: sertraline (Zoloft)

INTERVENTIONS:
Drug: sertraline (Zoloft) — Dosage form: Tablet, Dosage: over 25 mg/day, duration: Not defined

SUMMARY:
This is a multicenter retrospective study to investigate the dosage regimens of sertraline in the treatment of Posttraumatic Stress Disorder (PTSD) under current medical practice and the efficacy and safety of this drug in patients with PTSD. Data will be collected from the medical records of patients with PTSD.

DETAILED DESCRIPTION:
Patients with PTSD who have been dosed with sertraline from July 2006 (i.e., the start of marketing of this drug in Japan) or later to before contracting with each investigational site.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PTSD who have been dosed with sertraline since July 2006 or later.
* Patients must be Japanese.
* Patients should be started before the conclusion of a contract with each investigational site.

Exclusion Criteria:

* Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PTSD
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Japan (4):
  - KURUME University School of Medicine, Kurume, Fukuoka
  - Hyogo Institute for Traumatic Stress, Chuo-ku,Kobe-city, Hyōgo
  - National Defense Medical College/Department of Psychiatry, Tokorozawa, Saitama
  - Institute of Women?s Health Tokyo Women?s Medical University, Shinjyuku-ku, Tokyo

REFERENCES:
- [Derived] Kamo T, Maeda M, Oe M, Kato H, Shigemura J, Kuribayashi K, Hoshino Y. Dosage, effectiveness, and safety of sertraline treatment for posttraumatic stress disorder in a Japanese clinical setting: a retrospective study. BMC Psychiatry. 2016 Dec 7;16(1):434. doi: 10.1186/s12888-016-1138-5. PMID 27923359
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501099&StudyName=A%20Retrospective%20And%20Multicenter%20Survey%20To%20Investigate%20The%20Dosage%2C%20Efficacy%20And%20Safety%20Of%20Sertraline%20In%20Posttraumatic%20Stress%20Disorder%20Pat

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected from the medical records of participants with post-traumatic stress disorder (PTSD) who have been dosed with sertraline since July 2006 (i.e., the start of marketing of this drug in Japan) or later. Treatment with sertraline had to be initiated before the conclusion of the contract with investigational sites.
Pre-assignment Details: In this retrospective investigation, 123 patients were enrolled, but it was found during the data screening that one patient was not actually diagnosed with PTSD, and this patient was excluded from the investigation. Thus, 122 patients became subject to the investigation.
Groups:
- SERTRALINE: Participants with post-traumatic stress disorder (PTSD) who were treated with sertraline as instructed by physicians
Period: Overall Study
Arm/Group | SERTRALINE
Started | 122
Completed | 29
Not Completed | 93
Not completed — Adverse Event | 15
Not completed — Lack of Efficacy | 16
Not completed — Lost to Follow-up | 25
Not completed — Continuation | 33
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Groups:
- SERTRALINE: Participants with PTSD who were treated with sertraline as instructed by physicians.
Arm/Group | SERTRALINE
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 119
  MALE | 3

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression - Improvement (CGI-I) at End of Administration/Observation
Description: Number of participants in each category of CGI-I at end of administration/observation. CGI-I is a 7-point clinician-rated scale, ranging from (1) Very much improved, (2)Much improved, (3) Minimally improved, (4) No change, (5) Minimally worse, (6) Much worse, and (7) Very much worse.
Time Frame: Up to 6 years
Population: Full analysis set (FAS) was defined as those who had a record of either CGI-I or Clinical Global Impression of Severity (CGI-S).
Measure: Number; unit: Participants
Groups:
- Sertraline (Zoloft): Participants with PTSD who were treated with sertraline as instructed by physicians
Arm/Group | Sertraline (Zoloft)
Number analyzed (Participants) | 122
Participants
  Very much improved | 23
  Much improved | 38
  Minimally improved | 25
  No change | 32
  Minimally worse | 4
  Much worse | 0
  Very much worse | 0

2. Primary Outcome: Clinical Global Impression of Severity (CGI-S) at Start of Administration/Observation
Description: Number of participants in each category of CGI-S at start and end of administration/observation. CGI-S is a 7-point clinician-rated scale to assess severity of participant's current illness state, ranging from (1)Normal, not ill at all, (2)Borderline mentally ill, (3)Mildly ill, (4)Moderately ill, (5)Markedly ill, (6)Severely ill, (7)Among the most severely ill.
Time Frame: Start of administration
Population: FAS was defined as those who had a record of either CGI-I or CGI-S.
Measure: Number; unit: Participants
Arm/Group | Sertraline (Zoloft)
Number analyzed (Participants) | 122
Participants
  Normal at start | 0
  Borderline at start | 0
  Mild at start | 16
  Moderate at start | 68
  Marked at start | 17
  Severe at start | 20
  The most severe at start | 1

3. Primary Outcome: Clinical Global Impression of Severity (CGI-S) at End of Administration/Observation
Description: as for outcome 2
Time Frame: Up to 6 years
Population: FAS was defined as those who had a record of either CGI-I or CGI-S.
Measure: Number; unit: Participants
Arm/Group | Sertraline (Zoloft)
Number analyzed (Participants) | 122
Participants
  Normal at end | 13
  Borderline at end | 19
  Mild at end | 40
  Moderate at end | 40
  Marked at end | 4
  Severe at end | 5
  The most severe at end | 1

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | SERTRALINE
Serious Adverse Events (participants affected / at risk) | 7/122
Other Adverse Events (participants affected / at risk) | 71/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SERTRALINE (N=122)
Intentional overdose (Injury, poisoning and procedural complications) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hallucination (Psychiatric disorders) | 1
Intentional self-injury (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Thinking abnormal (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SERTRALINE (N=122)
Palpitations (Cardiac disorders) | 3
Hypoacusis (Ear and labyrinth disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Eye pain (Eye disorders) | 1
Photopsia (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Defaecation urgency (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 7
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 12
Stomatitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Feeling abnormal (General disorders) | 2
Inflammation (General disorders) | 1
Influenza like illness (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 4
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Seasonal allergy (Immune system disorders) | 1
Cystitis (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 4
Road traffic accident (Injury, poisoning and procedural complications) | 1
Blood cholesterol increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood prolactin increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Urine output decreased (Investigations) | 1
Weight increased (Investigations) | 2
White blood cell count increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyperphagia (Metabolism and nutrition disorders) | 4
Polydipsia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 12
Hypoaesthesia (Nervous system disorders) | 3
Sleep paralysis (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 11
Tremor (Nervous system disorders) | 3
Activation syndrome (Psychiatric disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Eating disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Intentional self-injury (Psychiatric disorders) | 2
Mania (Psychiatric disorders) | 1
Self injurious behaviour (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 1
Withdrawal syndrome (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Yawning (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.